CLINICAL TRIAL: NCT05528094
Title: An Exploratory Investigation of a Supplement to Support Student Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: JoySpring (Other)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20246
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Concentration Ability Impaired; Mental Fatigue
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GeniusDrops (Experimental): Once participants have signed the consent and assent, they will take the baseline survey to gather information about their ability to focus and concentration.
  Once in the study, participants will be asked to take two dropperfuls of the test product (Genius Drops) twice daily. The participants can take the dropperful directly or add it to drinks/snacks. Participants will need to be in school during the entirety of the study.
  Participants will take a subsequent survey after two weeks in the trial and then another survey at the end of the trial.
  Interventions: Dietary Supplement: GeniusDrops

INTERVENTIONS:
Dietary Supplement: GeniusDrops — The active ingredients listed below are safe and the study sponsor has noted there are no known side effects of the supplement. The main ingredients are:
  Hibiscus flower- Has been shown to boost oxygenation to the brain and vital organs. Has also demonstrated efficacy for boosting the immune system.
  Gingko leaf- Has been shown to stimulate memory by increasing mental sharpness and clarity.
  Rhodiola- Helps regulate energy and stress level. Gotu kola- Has been shown to have impacts on reducing anxiety. Licorice Root- Helps boost the key brain neurotransmitter called Brain Derived Neurotrophic factor which can help with cognitive development Peppermint Leaf- Reduces fatigue while helping improve cognitive abilities. Has also been shown to promote immune system function.

SUMMARY:
In this trial, the herbal supplement (GeniusDrops) will be tested to see the effects it has on the dependent variables of interest. Participants will take the supplement twice a day for a month and respond to surveys at study baseline, midpoint, and the conclusion of the study. The findings of this study will be used for marketing materials and to inform future trials using the supplement.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form and a parental assent form
* Must be experiencing issues with focus, mood, and memory
* Must be looking to improve classroom performance
* Gets easily distracted

Exclusion Criteria:

* Diagnosis of ADD or ADHD
* Currently taking a prescription medication meant to treat ADD or ADHD
* Diagnosed with additional conditions that would not allow them to adhere to the protocol.
* Willing to take a supplement targeting improving mood, concentration, and focus

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2022-04-14 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Examination of self-reported focus | 4 weeks
  Participants will respond to a survey to assess perceived changes in focus.
Examination of Self-reported concentration | 4 weeks
  Participants will respond to a survey to assess perceived changes in concentration
Examination of Self-reported mood states | 4 weeks
  Participants will respond to a survey to assess perceived changes in moods.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hill, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided